

# A two-year Clinical Impact of Bulk-fill Lowviscosity Resin Composite Liners in Class II Restorations

Local ethics committee approval number: M 11120520

Study Start: January 15, 2020 [Actual]

Primary Completion: April 27, 2022 [Actual]

Study Completion: June 17, 2023 [Actual]

By

# Mustafa Ahmed Alsharkawy, B. Dent, MSCD

Assistant Lecturer, Operative Dentistry Department
Faculty of Dentistry Mansoura University

### **Protocol:**

### Introduction

Patients' increasing desire for aesthetic restorations has led to the use of direct resin composites as the most versatile restoration for both anterior and posterior teeth, with evidence for their success.<sup>1-5</sup> However, polymerization shrinkage and indeed the strains it generates are still one of the main reasons for resin composite restoration failures. This is because it applies tension to the tooth-restoration interface over time, endangering the bonding integrity.<sup>6</sup> Furthermore, these stresses negatively affect cavity margins with leakage and subsequent carious lesion development.<sup>7</sup>

These stresses are widely recognized to be affected by the placement techniques.<sup>8</sup> The standard method for avoiding the clinical effects of polymerization stress is incremental layering.<sup>9-13</sup> The drawbacks of this technique are the possibilities of voids or contaminants inclusion between layers, and difficulties in filling conservative cavities.<sup>14-16</sup> In addition to, a need for restorative procedures that effectively shorten restoration time. In this regard, bulk-fill high-viscosity(regular), and low-viscosity (flowable) methacrylate-based resin composites had been evolved.<sup>17-21</sup>

Different viscosities are due to filler content that has direct relation with material modulus of elasticity.<sup>22</sup> Bulk-fill low-viscosity resin composites (BLRC) are indicated as liners and stress absorbers in class I and class II cavities, requiring an additional layer high-viscosity type.<sup>23</sup> 10, 24-26 While high viscosity (BHRC) types can be inserted up to 5 mm increment, without the need of a veneering layer. <sup>27-30</sup> The increased curing depth were attributed to monomers which act as modulators in the polymerization reaction, resulting in reduced shrinkage.<sup>31-35</sup>

Scientific evidence has shown that bulk-fill resin composites have comparable polymerization shrinkage and stress, depth of cure, physic mechanical properties, and marginal adaptation when compared to conventional composites. <sup>15,</sup> <sup>34-41</sup> Other studies have revealed greater values for shrinkage vectors and a higher tendency for debonding. <sup>42</sup> In relation to their clinical performance, data investigating the high-viscosity methacrylate based types had a heterogeneous behaviour and depended mainly in their chemical composition. <sup>43-45</sup> <sup>46, 47</sup> Most of the studies have reported similar results related to marginal degradation when compared to conventional resin composites. <sup>46, 48</sup>

Bulk-fill low-viscosity resin composites (BLRC) as liners demonstrated a stress reduction ability in posterior resin composite restorations, thereby exhibiting a high level of clinical efficacy over three years evaluation. <sup>23, 49-54</sup> Besides, their low elastic modulus may provide a certain stress-absorbing layer, thus relieving the polymerization stress of the veneering regular viscosity composites. <sup>55-58, 14</sup> Moreover, subsequent layer of higher modulus resin composites can be absorbed by an elastic intermediary layer, lowering stress at the tooth-restoration interface. In a RCT one of the restorative systems that used BLRC liner showed the lowest surface staining. <sup>54</sup>

Despite, contradictory evidence had reported decreased adaption and higher polymerization shrinkage stress than the high-viscosity counterpart and other study found no improvement in the clinical performance of a class II restoration .<sup>59, 60</sup> It is unknown, nevertheless, whether low viscosity bulk-fill composites would be susceptible to proximal contact defects comparable to those reported in glass ionomer restoratives.<sup>61, 62</sup>

Resin matrix plays an important role on the shrinkage behaviour of resin composite restorations.<sup>63</sup> The high molecular weight bis-GMA (bisphenol A-glycidyl methacrylate) has been the main monomer used in methacrylate-based resin composites since their development.<sup>64</sup> Due to the high viscosity of this monomer, low molecular weight monomers (diluents) were added to the final blend to get a suitable formulation for clinical use and to allow filler inclusion.<sup>65</sup> These diluent monomers were supposed to increase the polymerization shrinkage of resin composites.<sup>66</sup>

To reduce the clinical problems associated with the conventional methacrylate based resin composites, Ormocers were developed.<sup>67-71</sup> They claimed to lower polymerization stress due to their reduced amount of organic resin.<sup>67, 69, 72-76</sup> On the other hand, their first launched generations did not make any clear progress over the methacrylate-based resin composites.<sup>77</sup> A probable explanation of the attained findings was the inclusion of methacrylate monomers beside ormocer molecule that served as diluents.<sup>78</sup> A pure ormocer resin composite was then introduced to the market and it was placed by incremental layering.<sup>75, 76, 79</sup>

In addition to layering method, the pure material had been implemented for bulk-filling with two viscosities like methacrylates (high viscosity, low viscosity). In comparison with methacrylate resin composites, the pure ormocer material were supposed to lower polymerization shrinkage.<sup>75, 76</sup> Bulk-fill high-viscosity ormocer-based resin composites(BHORC) may be superior alternative to the standard layering method, given similar clinical performance after 24 months, with the advantage of simplified procedures.<sup>80</sup> In addition, a RCT utilized the pure layered ormocer material (Admira-fusion) and found non-significant differences over the compared methacrylate based resin composites after 24 months in class II restorations.<sup>79</sup>

As regard lining ormocer-based resin composites, the data is scarce. Torres et al<sup>81</sup> reported in a one randomized clinical trial to have no influence in their clinical performance. So that the aim of this randomized, split-mouth clinical trial was to evaluate the clinical performance of class II restorations made with the use of BHORC versus BHMRC composites either placed alone or with the effect of BLRC liner of the same type after 2 years follow up.

The null hypotheses in the study were as follows: (1) Different types of matrix structures (ormocer vs. methacrylate) have no effect on the clinical performance of restorations; (2) A layer of bulk-fill resin composite liner of the same category would not affect clinical parameters evaluated.

# Aim of the study

The current study was intended to evaluate the effect of flowable lining resin composites on 2-year clinical performance of bulk-fill ormocer versus methacrylate-based restorative systems in class II cavities according to FDI criteria.

# **Null hypothesis**

The null hypothesis that will be tested in this project is that there would be no significant difference among the four tested restorative strategies at different clinical evaluation periods.

#### **Materials and Methods**

#### **Materials**

Bulk-fill high viscosity methacrylate-based resin composite (BHMRC) (XTra-fill Voco, Germany), Bulk-fill high-viscosity ormocer-based resin composite (BHORC) (Admira-Fusion-Xtra Voco, Germany), Bulk-fill low-viscosity methacrylate-based resin composite (XTra-Base Voco, Germany) (BLMRC) and bulk-fill low-viscosity ormocer-based resin composite (BLORC) (Admira-Fusion-Base Voco, Germany). All restorations were performed using the universal adhesive (Futura U bond Voco, Germany).

#### Methods

# Clinical trial design

This clinical trial will be conducted according to CONSORT guidelines for Randomized Clinical Trials (RCTs).<sup>45</sup> It will be carried out after gaining approval from Medical Ethics Committee of Mansoura University.

#### Recruitment

Patients enrolled in this study were from the Outpatient Clinic at Mansoura University, Faculty of Dentistry. Patients were informed on the background of the study and who accepted the study condition signed a consent form. The consent form was approved by the ethical committee at faculty of dentistry, Mansoura University.

# Eligibility criteria

Participants were examined to form a group with 30 patients that justify the inclusion and exclusion criteria. Patients were required to have good general health, be older than 18 years old. Patients with extremely poor oral hygiene, severe or chronic periodontitis, or heavy bruxism habits will be excluded from the study.

Patients had to present at least four teeth with class II cavities to be restored (molars or premolar). Also, unsatisfactory class II restorations that are moderately deep with an adjacent tooth was involved.

#### Randomization

Randomization was applied by noting each tooth to be restored (FDI 2- digit code) on one paper and type of restorative strategy on a second. First, a tooth number was drawn blindly. Subsequently a restorative protocol was allocated to this tooth by blind drawing. This procedure was repeated if more than three restorations must be placed.

### **Interventions: Restorative procedures**

A split-mouth design was used in this study. For ormocer- based resin composite restorative system, it will be placed without resin flowable liner in one side, while it will be lined in the other side. The same protocol will be applied for methacrylate-based resin composite restorative system. Hence, each patient will receive four restorations with different strategies. All restorative procedures will be carried out by a single operator.

After administration of local anesthetic, rubber dam will be placed. The cavity preparation was then carried out with an outline limited to caries progression. The cavities depth in mm will be measured by a periodontal probe to give an idea about the thickness of the flowable composite liner (when used) and preserve 2 mm depth for the overlying resin. Restorative systems were then be applied according to the instructions recommended by their manufactures. Sectional pre-contoured matrix with ring, and wave like contour plastic wedges was used to restore the shape of the proximal walls. Adhesive and resin composites was cured using a LED (light

emitting diode) curing unit in the standard application mode and an output of  $650 \, \text{mW/cm}^2$ .

### **Clinical evaluation**

All restorations were clinically evaluated using FDI criteria.<sup>46</sup> This evaluation was done at the baseline, then after 12-month and finally at 24-months.

# Statistical analysis:

The Chi-Square test was used for comparison between the four groups within every follow up period, while marginal homogeneity test was used to compare the changes within each group per time.

# **Results:**

Table: Scores of all tested criteria and results of Chi-Square and Marginal homogeneity tests

| category | | eline<br>=30) | # | 6 Months<br>(n=30) # | | | | | Mont | | | # | 18 Months<br>(n=30) | | | | 24 Months<br># (n=30) | | | | # | XF s | XB s | AFX <sup>8</sup> | AFB § | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| category | | KB AFX AFB | " | | XB AF | AFB | Ι ″ | | XB | | AFB | " | | | AFX A | FB | " | | | AFX | AFB | " | 241 | AD | ALIZ | AFD |
| | | 30 30 30 | | 30 | 30 30 | | | 30 | 30 | | 30 | | 30 | 30 | 30 | 30 | p=1.0 | 30 | 30 | 30 | 30 | | p1=1.0 | p1=1.0 | p1=1.0 | p1=1.0 |
| | 2 0 | 0 0 0 | | 0 | 0 0 | 0 | 0 <b>p=1.0</b> | 0 | 0 | 0 | 0 | p=1.0 | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | p2=1.0 | p2=1.0 | p2=1.0 | p2=1.0 |
| Marginal staining | 3 0 | 0 0 0 | p=1.0 | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 p | | 0 | 0 | 0 | 0 | p=1.0 | p3=1.0 | p3=1.0 | p3=1.0 | p3=1.0 |
| | 4 0 | 0 0 0 | - | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | p4=1.0 | p4=1.0 | p4=1.0 | p4=1.0 |
| | 5 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | | | | |
| | 1 28 1 | 29 30 30 | | 28 | 29 30 | 30 | | 28 | 29 | 30 | 30 | | 28 | 29 | 30 | 30 | | 28 | 29 | 30 | 30 | | p1=1.0 | p1=1.0 | p1=1.0 | p1=1.0 |
| | 2 2 | 1 0 0 | | 2 | 1 0 | 0 | | 2 | 1 | 0 | 0 | | 2 | 1 | 0 | 0 | | 2 | 1 | 0 | 0 | | p2=1.0 | p2=1.0 | p2=1.0 | p2=1.0 |
| Color match and translucency | 3 0 | 0 0 0 | p=0.288 | 0 | 0 0 | 0 | p=0.288 | 0 | 0 | 0 | 0 | p=0.288 | 0 | 0 | 0 | 0 <b>p</b> = | p=0.288 | 0 | 0 | 0 | 0 | p=0.288 | p3=1.0 | p3=1.0 | p3=1.0 | p3=1.0 |
| | 4 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | p4=1.0 | p4=1.0 | p4=1.0 | p4=1.0 |
| | 5 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | | | | |
| | 1 30 3 | 30 30 30 | | 30 | 30 30 | 30 | | 30 | 30 | 30 | 30 | p=1.0 | 30 | 30 | 30 | 30 | | 30 | 30 | 30 | 30 | | p1=1.0 | p1=1.0 | p1=1.0 | p1=1.0 |
| Fracture of material and | 2 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | p2=1.0 | p2=1.0 | p2=1.0 | p2=1.0 |
| retention | 3 0 | 0 0 0 | p=1.0 | 0 | 0 0 | 0 | p=1.0 | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 p | p=1.0 | 0 | 0 | 0 | 0 | p=1.0 | p3=1.0 | p3=1.0 | p3=1.0 | p3=1.0 |
| | 4 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | p4=1.0 | p4=1.0 | p4=1.0 | p4=1.0 |
| | 5 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | | | | |
| Marginal adaptation | 1 30 3 | 30 30 30 | | 30 | 30 30 | 30 | | 30 | 30 | 30 | 30 | p=1.0 | 30 | 30 | 30 | 30 | p=1.0 | 30 | 30 | 30 | 30 | p=1.0 | p1=1.0 | p1=1.0 | p1=1.0 | p1=1.0 |
| | 2 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | p2=1.0 | p2=1.0 | p2=1.0 | p2=1.0 |
| | 3 0 | 0 0 0 | p=1.0 | 0 | 0 0 | 0 | p=1.0 | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 p | | 0 | 0 | 0 | 0 | | p3=1.0 | p3=1.0 | p3=1.0 | p3=1.0 |
| | 4 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | p4=1.0 | p4=1.0 | p4=1.0 | p4=1.0 |
| | 5 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 0 0 | | 0 | 0 | 0 | 0 | | | | | | | |
| | | 30 30 30 | | 30 | 30 30 | 30 | | 30 | 30 | 30 | 30 | p=1.0 | 30 | 30 | | 30 | p=1.0 | 30 | 30 | 30 | 30 | | p1=1.0 | p1=1.0 | p1=1.0 | p1=1.0 |
| | 2 0 | 0 0 0 | p=1.0 | 0 | 0 0 | 0 | p=1.0 | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | p2=1.0 | p2=1.0 | p2=1.0 | p2=1.0 |
| Radiographic examination | 3 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | | _ | | 0 | 0 | 0 | 0 | p=1.0 | p3=1.0 | p3=1.0 | p3=1.0 | p3=1.0 |
| | 4 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | | 0 | | 0 | 0 | 0 | 0 | | p4=1.0 | p4=1.0 | p4=1.0 | p4=1.0 |
| | 5 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | | 0 | | 0 | 0 | 0 | 0 | | | | | |
| | | 30 30 30 | | 30 | 30 30 | 30 | | 30 | 30 | | 30 | | 30 | 30 | | 30 | | 29 | 28 | 27 | 28 | | <b>p1</b> =0.317 | | | - |
| | _ ` | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | | 0 | | 1 | 2 | 3 | 2 | | | p2=0.157 | _ | - |
| Interproximal contact | | 0 0 0 | p=1.0 | 0 | 0 0 | 0 | p=1.0 | 0 0 0 | 0 <b>p=1</b> | p=1.0 | 0 | 0 | - | _ | p=1.0 | 0 | 0 | 0 | 0 | p=0.784 | | p3=0.083 | | | | |
| | | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 0 0 0 | | | 0 | 0 | | 0 | | 0 | 0 | 0 | 0 | | p4=0.157 | p4=0.157 | p4=0.157 | p4=0.157 | |
| | | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | | 0 | | 0 | 0 | 0 | 0 | | | | | |
| | | 30 28 30 | | 30 | 30 30 | 30 | | 30 | 30 | | 30 | | 30 | 30 | | 30 | p=1.0 | 30 | 30 | 30 | 30 | | p1=0.317 | p1=0.157 | p1=0.083 | - |
| Postoperative (hyper-) | _ | 0 2 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | - | 0 | | 0 | 0 | 0 | 0 | p=1.0 | p2=1.0 | p2=1.0 | p2=1.0 | p2=1.0 |
| sensitivity and tooth vitality | _ | 0 0 0 | p=0.288 | 0 | 0 0 | 0 | p=1.0 | 0 | 0 | 0 | 0 | p=1.0 | 0 | 0 | | | | 0 | 0 | 0 | 0 | | p3=0.157 | p3=0.157 | p3=0.157 | 1 |
| | | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | | 0 | | 0 | 0 | 0 | 0 | | p4=1.0 | p4=1.0 | p4=1.0 | p4=1.0 |
| | J . | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 0 0 | | | 0 | 0 | 0 | 0 | | | | | | |
| | | 30 30 30 | | 30 | 30 30 | | | 30 | 30 | 30 | 30 | | 30 | 30 | 30 | _ | | 30 | 30 | 30 | 30 | | p1=1.0 | p1=1.0 | p1=1.0 | p1=1.0 |
| Recurrent caries | | 0 0 0 | p=1.0 | 0 | 0 0 | 0 | p=1.0 | 0 | 0 | 0 | 0 | p=1.0 | 0 | 0 | | - | p=1.0 | 0 | 0 | 0 | 0 | p=1.0 | p2=1.0 | p2=1.0 | p2=1.0 | p2=1.0 |
| | 3 0 | 0 0 0 | | 0 | 0 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | p3=1.0 | p3=1.0 | p3=1.0 | p3=1.0 |

| | 4 | 0 | 0 | 0 | ) | 0 | | 0 | 0 | 0 | 0 0 | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 0 | 0 | 0 | | p4=1.0 | p4=1.0 | p4=1.0 | p4=1.0 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 5 | 0 | 0 | 0 | ) | 0 | | 0 | 0 | 0 | 0 | | 0 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | | | | |
| Tooth integrity (enamel cracks and tooth fractures) | 1 | 30 | 30 | 30 | 0 : | 30 | p=1.0 | 30 | 30 | 30 | 30 | _ | 30 | 30 | 30 | 30 | 0<br>0 <b>p=1.0</b> | 30 | 30 | 30 | 30 | p=1.0 | 30 | 30 | 30 | 30 | | p1=1.0 | p1=1.0 | p1=1.0 | p1=1.0 |
| | 2 | 0 | 0 | 0 | ) | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 ( | 0 | 0 | | p2=1.0 | p2=1.0 | p2=1.0 | p2=1.0 |
| | 3 | 0 | 0 | 0 | ) | 0 | | 0 | 0 | 0 | 0 | p=1.0 | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | p=1.0 | | p3=1.0 | p3=1.0 | p3=1.0 |
| | 4 | 0 | 0 | 0 | ) | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | p4=1.0 | p4=1.0 | p4=1.0 | p4=1.0 |
| | 5 | 0 | 0 | 0 | ) | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | 0 | 0 | 0 | 0 | | | | | |

#USED test: Chi-Square test for comparing between groups (EXF, SDR and TNFBF) \$USED test: Marginal Homogeneity test for comparing between different follow up times as compared to baseline value

#### **References:**

- 1. Lynch C, Opdam N, Hickel R, Brunton P, Gurgan S, Kakaboura A, et al. Academy of Operative Dentistry European Section: guidance on the use of resin composites for direct restoration of posterior teeth. J Dent. 2014;42:377-83.
- 2. Sunnegårdh-Grönberg K, van Dijken JW, Funegård U, Lindberg A, Nilsson M. Selection of dental materials and longevity of replaced restorations in Public Dental Health clinics in northern Sweden. J Dent. 2009;37:673-8.
- 3. Ástvaldsdóttir Á, Dagerhamn J, van Dijken JW, Naimi-Akbar A, Sandborgh-Englund G, Tranaeus S, et al. Longevity of posterior resin composite restorations in adults–A systematic review. J Dent. 2015;43:934-54.
- 4. De Andrade A, Duarte R, Silva FMe, Batista A, Lima K, Monteiro G, et al. Resin composite class I restorations: a 54-month randomized clinical trial. Oper Dent. 2014;39:588-94.
- **5.** Opdam N. Sande FH van de, Bronkhorst E, et al. Longevity of posterior composite restorations: a systematic review and meta-analysis. J Dent Res. 2014; 93:943-9.
- 6. Schmidt M, Dige I, Kirkevang L-L, Vaeth M, Hørsted-Bindslev P. Five-year evaluation of a low-shrinkage Silorane resin composite material: a randomized clinical trial. Clin Oral Investig. 2015;19:245-51.

- 7. Van Dijken JW, Pallesen U. A six-year prospective randomized study of a nanohybrid and a conventional hybrid resin composite in class II restorations. Dent Mater. 2013;29:191-8.
- 8. Gomes I, Mariz D, Borges A, Tonetto M, Firoozmand L, Kuga C, et al. In vivo evaluation of proximal resin composite restorations performed using three different matrix systems. J Contemp Dent Pract. 2015;16:643-7.
- 9. El-Shamy H, Saber M, Dörfer C, El-Badrawy W, Loomans B. Influence of volumetric shrinkage and curing light intensity on proximal contact tightness of class II resin composite restorations: in vitro study. Oper Dent. 2012;37:205-10.
- 10. Braga RR, Ballester RY, Ferracane JL. Factors involved in the development of polymerization shrinkage stress in resin-composites: a systematic review. Dent Mater. 2005;21:962-70.
- 11. Van Dijken JW, Pallesen U. A randomized controlled three year evaluation of "bulk-filled" posterior resin restorations based on stress decreasing resin technology. Dent Mater. 2014;30:e245-e51.
- 12. Van Dijken JW, Pallesen U. Bulk-filled posterior resin restorations based on stress-decreasing resin technology: a randomized, controlled 6-year evaluation. Eur J Oral Sci. 2017;125:303-9.
- 13. Veloso SRM, Lemos CAA, de Moraes SLD, do Egito Vasconcelos BC, Pellizzer EP, de Melo Monteiro GQ. Clinical performance of bulk-fill and conventional resin

composite restorations in posterior teeth: a systematic review and meta-analysis. Clin Oral Investig. 2019;23:221-33.

- 14. Ferracane J, Berge H, Condon J. In vitro aging of dental composites in water—effect of degree of conversion, filler volume, and filler/matrix coupling. J Biomed Mater Res. 1998;42:465-72.
- 15. Weinmann W, Thalacker C, Guggenberger R. Siloranes in dental composites. Dent Mater. 2005;21:68-74.
- 16. Frascino S, Fagundes T, Silva U, Rahal V, Barboza A, Santos P, et al. Randomized prospective clinical trial of class II restorations using low-shrinkage flowable resin composite. Oper Dent. 2019.
- 17. Cakir D, Sergent R, Burgess JO. Polymerization shrinkage—A clinical review. Inside Dent. 2007;3:3-10.
- 18. Manhart J. Nanohybrid-ORMOCER®-Füllungsmaterial für die Bulk-Fill-Technik. Stomatologie. 2015;112:266-7.
- 19. Kalra S, Singh A, Gupta M, Chadha V. Ormocer: an aesthetic direct restorative material; an in vitro study comparing the marginal sealing ability of organically modified ceramics and a hybrid composite using an ormocer-based bonding agent and a conventional fifth-generation bonding agent. Contemp Clin Dent. 2012;3:48.
- 20. Marghalani HY, Watts DC. Viscoelastic stability of resin-composites aged in food-simulating solvents. Dent Mater. 2013;29:963-70.

- 21. Shafqat SS, Hamdan S, Rigit ARH, Tien NKH, Saleh SF, Khan AA, editors. Synthesis and characterization of heterocyclic-ORMOCERS composites through Sol-gel process: a review. 5th International Conference on Science & Technology: Applications in Industry & Education (ICSTIE 2014).
- 22. Bottenberg P, Alaerts M, Keulemans F. A prospective randomised clinical trial of one bis-GMA-based and two ormocer-based composite restorative systems in class II cavities: three-year results. J Dent. 2007;35:163-71.
- 23. Bottenberg P, Jacquet W, Alaerts M, Keulemans F. A prospective randomized clinical trial of one bis-GMA-based and two ormocer-based composite restorative systems in class II cavities: Five-year results. J Dent. 2009;37:198-203.
- 24. Monsarrat P, Garnier S, Vergnes J-N, Nasr K, Grosgogeat B, Joniot S. Survival of directly placed ormocer-based restorative materials: A systematic review and meta-analysis of clinical trials. Dent Mater. 2017;33:e212-e20.
- 25. Klauer E, Belli R, Petschelt A, Lohbauer U. Mechanical and hydrolytic degradation of an Ormocer®-based Bis-GMA-free resin composite. Clin Oral Investig. 2019;23:2113-21.
- 26. Klauer E, Belli R, Petschelt A, Lohbauer U. Mechanical and hydrolytic degradation of an Ormocer®-based Bis-GMA-free resin composite. Clin Oral Investig. 2019;23:2113-21.

- 27. Carvalho RMd, Pereira JC, Yoshiyama M, Pashley DH. A review of polymerization contraction: The influence of stress development versus stress relief. Oper Dent. 1996;21:17-24.
- 28. Kleverlaan CJ, Feilzer AJ. Polymerization shrinkage and contraction stress of dental resin composites. Dent Mater. 2005;21:1150-7.
- 29. Ferracane J. Placing dental composites—a stressful experience. Oper Dent. 2008;33:247-57.
- 30. Abbas G, Fleming G, Harrington E, Shortall A, Burke F. Cuspal movement and microleakage in premolar teeth restored with a packable composite cured in bulk or in increments. J Dent. 2003;31:437-44.
- 31. Lazarchik DA, Hammond BD, Sikes CL, Looney SW, Rueggeberg FA. Hardness comparison of bulk-filled/transtooth and incremental-filled/occlusally irradiated composite resins. J Prosthet Dent 2007;98:129-40.
- 32. Alrahlah A, Silikas N, Watts D. Post-cure depth of cure of bulk fill dental resincomposites. Dent Mater. 2014;30:149-54.
- 33. Ilie N, Keßler A, Durner J. Influence of various irradiation processes on the mechanical properties and polymerisation kinetics of bulk-fill resin based composites. J Dent. 2013;41:695-702.

- 34. Tarle Z, Attin T, Marovic D, Andermatt L, Ristic M, Tauböck TT. Influence of irradiation time on subsurface degree of conversion and microhardness of high-viscosity bulk-fill resin composites. Clin Oral Investig. 2015;19:831-40.
- 35. Tauböck TT, Marovic D, Zeljezic D, Steingruber AD, Attin T, Tarle Z. Genotoxic potential of dental bulk-fill resin composites. Dent Mater. 2017;33:788-95.
- 36. Ólafsson VG, Ritter AV, Swift Jr EJ, Boushell LW, Ko CC, Jackson GR, et al. Effect of composite type and placement technique on cuspal strain. J Esthet Restor Dent. 2018;30:30-8.
- 37. Rosatto C, Bicalho A, Veríssimo C, Bragança G, Rodrigues M, Tantbirojn D, et al. Mechanical properties, shrinkage stress, cuspal strain and fracture resistance of molars restored with bulk-fill composites and incremental filling technique. J Dent. 2015;43:1519-28.
- 38. Yazici A, Antonson S, Kutuk Z, Ergin E. Thirty-six-month clinical comparison of bulk fill and nanofill composite restorations. OPer Dent. 2017;42:478-85.
- 39. Hickey D, Sharif O, Janjua F, Brunton P. Bulk dentine replacement versus incrementally placed resin composite: A randomised controlled clinical trial. J Dent. 2016;46:18-22.

- 40. Boaro LCC, Lopes DP, de Souza ASC, Nakano EL, Perez MDA, Pfeifer CS, et al. Clinical performance and chemical-physical properties of bulk fill composites resin—a systematic review and meta-analysis. Dent Mater. 2019.
- 41. Tauböck TT, Jäger F, Attin T. Polymerization shrinkage and shrinkage force kinetics of high-and low-viscosity dimethacrylate-and ormocer-based bulk-fill resin composites. Odontology. 2019;107:103-10.
- 42. Sadeghi M, Lynch C. The effect of flowable materials on the microleakage of class II composite restorations that extend apical to the cemento-enamel junction. Oper Dent. 2009;34:306-11.
- 43. Bakhsh TA, Sadr A, Shimada Y, Turkistani A, Abuljadayel R, Tagami J. Does lining class-II cavities with flowable composite improve the interfacial adaptation? J ADHES SCI TECHNOL. 2019:1-17.
- 44. Oglakci B, Kazak M, Donmez N, Dalkilic EE, Koymen SS. The use of a liner under different bulk-fill resin composites: 3D GAP formation analysis by x-ray microcomputed tomography. J Appl Oral Sci. 2020;28.
- 45. Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. BMC medicine. 2010;8:18.
- 46. Hickel R, Peschke A, Tyas M, Mjör I, Bayne S, Peters M, et al. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations—update and clinical examples. Clin Oral Investig. 2010;14:349-66.